CLINICAL TRIAL: NCT00874653
Title: Levonorgestrel Releasing Intrauterine System (MIRENA) in Idiopathic Menorrhagia
Brief Title: Survey on Patient Satisfaction Rate for Mirena Use in Heavy Menstrual Bleeding
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14175; MA0711IT (Other: Other company ID)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levonorgestrel (Mirena, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel (Mirena, BAY86-5028) — Women using Mirena for intrauterine treatment of menorrhagia

SUMMARY:
The purposes of this study are:

* To evaluate patient satisfaction for efficacy and tolerability of heavy menstrual bleeding treatment by Mirena.
* To collect italian data for Mirena in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Idiopathic Menorrhagia and Mirena inserted for a period no longer than three months according to the assessment of the investigator and according to the international and national guidelines. These women should also accept to be on contraception during the time period that they have Mirena in situ
* Body Mass Index = 18-30

Exclusion Criteria:

* One or more of the following disorders: Current or recurrent pelvic inflammatory disease; infection of the lower genital tract; postpartum endometritis; septic abortion during the past three months; cervicitis; cervical dysplasia; uterine or cervical malignancy; undiagnosed abnormal uterine bleeding; congenital or acquired abnormality of the uterus including fibroids if they distort the uterine cavity; conditions associated with increased susceptibility to infections; acute liver disease or liver tumor; known hypersensitivity to any of the constituents of the product
* Nulliparity
* Consumption of Iron, Antiprostaglandins, hormonal drugs and any medication that could effect bleeding should be stopped at least 3 months before the first visit and should not be used during the course of the study.
* History of diabetes mellitus, cardiovascular disease and thyroid abnormalities
* Anticoagulation therapy
* Cancer history including breast cancer

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with a diagnosis of idiopathic menorrhagia and Mirena inserted for a period no longer than three months according to the assessment of the investigator will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2008-04; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The quality of life on the basis of the validated Health-Related Quality of Life questionnaire (HRQL SF-36) | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Italy